CLINICAL TRIAL: NCT01592721
Title: Safety and Efficacy of Radiation and Cetuximab Plus Intratumoral EGFR Antisense DNA in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Radiation and Cetuximab Plus Intratumoral EGFR Antisense DNA in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRC 11-47; HSC20120131H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-04-26; First posted 2012-05-07 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: Carcinoma; Squamous cell carcinoma; Head and neck neoplasms; Cetuximab
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGFR Antisense DNA (Experimental): EGFR AS will be administered by direct intratumoral injection using direct visualization, endoscopy, or imaging-guidance (ultrasound) as clinically determined. Patients will receive a total of up to 4 weekly intratumoral injections of EGFR antisense (or less if there is no identifiable tumor) starting 2 weeks prior to radiation. Patients will receive standard radiation 70 Gy/200 cGy/daily, 5 days/week, with concurrent cetuximab 250 mg/m2, after a loading dose of 400 mg/m2 2 weeks prior to starting radiation.
  Interventions: Biological: EGFR Antisense DNA

INTERVENTIONS:
Biological: EGFR Antisense DNA — EGFR AS will be administered by direct intratumoral injection using direct visualization, endoscopy, or imaging-guidance (ultrasound) as clinically determined. Patients will receive a total of up to 4 weekly intratumoral injections of EGFR antisense (or less if there is no identifiable tumor) starting 2 weeks prior to radiation. Patients will receive standard radiation 70 Gy/200 cGy/daily, 5 days/week, with concurrent cetuximab 250 mg/m2, after a loading dose of 400 mg/m2 2 weeks prior to starting radiation.

SUMMARY:
The incorporation of novel targeted therapies to radiation therapy is of particular interest in head and neck cancer and may improve efficacy without significantly increasing toxicity. The investigators hypothesize that the addition of a second EGFR-targeted agent that inhibits EGFR at the intracellular level will improve the antitumor effect of standard radiation and cetuximab. The goal of this study is to evaluate the safety, efficacy, and the biologic effects in patients with locally advanced SCCHN of an antisense gene targeting the EGFR in combination with standard therapy with radiation and cetuximab.

DETAILED DESCRIPTION:
The Epidermal Growth Factor Receptor (EGFR) is highly expressed in SCCHN and its overexpression is associated with poor patient outcome. EGFR is a promising target of anticancer therapy. The investigators have developed EGFR antisense DNA as a safe and potentially efficacious treatment for SCCHN as shown in a previous phase I study conducted at the University of Pittsburgh. Cetuximab (Erbitux or C225) is a chimerized EGFR monoclonal antibody that has produced positive results in a phase III trial in SCCHN when added to radiation therapy and was approved by the FDA for the treatment of locally advanced SCCHN. Radiation plus cetuximab is considered a standard treatment, especially for patients who are not good candidates for chemotherapy. In the current study, the investigators plan to evaluate the addition of intratumoral EGFR antisense DNA (EGFR AS) to standard radiation with concurrent cetuximab in patients.

Objectives

* To evaluate the safety of the combination of intratumoral EGFS AS DNA with standard cetuximab and radiation.
* To evaluate the locoregional progression-free survival in selected patients with locally advanced SCCHN treated with intratumoral EGFR AS DNA combined with standard radiation plus cetuximab.
* To evaluate other efficacy parameters, including the objective response rate, distant control and overall progression-free survival, and overall survival.
* To determine the effect of EGFR antisense therapy on EGFR-related biomarkers. The investigators will use reverse phase protein microarrays (RPPA) and immunohistochemical (IHC) analysis of tissue microarrays (TMA) on baseline and post-treatment tumor tissue to determine the expression level and modulation of a panel of EGFR and EGFR-pathway related biomarkers, including (but not necessarily limited to) EGFR, pEGFR, Src, pMAPK, STAT3, pSTAT3, pSTAT5, pSTAT1, pAKT, p38, p21, p27, PARP, E-cadherin, p-ErbB3, and Ki67.
* To examine the transfection of the EGFR antisense gene therapy in vivo.

Subject population

The investigators will enroll patients with SCCHN who are suitable for intratumoral injections of EGFR antisense.

Treatment plan

EGFR AS will be administered by direct intratumoral injection using direct visualization, endoscopy, or imaging-guidance (ultrasound) as clinically determined (see protocol). Patients will receive a total of up to 4 weekly intratumoral injections of EGFR antisense (or less if there is no identifiable tumor) starting 2 weeks prior to radiation (study schema in protocol). Patients will receive standard radiation 70 Gy/200 cGy/daily, 5 days/week, with concurrent cetuximab 250 mg/m2, after a loading dose of 400 mg/m2 2 weeks prior to starting radiation.

Statistical Design and Sample Size

The study will be conducted in two-stages. In the first stage, 11 patients with stage IVA-C or recurrent disease will be evaluated for safety. If the regimen is deemed safe, a total of 31 patients with stage III or IVA-B, previously untreated SCCHN will be enrolled in the second stage of the study.

ELIGIBILITY:
Inclusion Criteria:

* First stage Patients with AJCC 7th edition stage IVA-IVC or recurrent or metastatic head and neck cancer will be eligible. Patients with M1 disease must have asymptomatic or low volume distant metastasis and require palliation for local and regional disease.
* Second stage (phase II part) Patients with AJCC 7th edition stage III-IVB (T1-T4, N1-3M0) head and neck cancer, except WHO type II and III nasopharyngeal cancer, including unknown primary tumors.
* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma or variants or poorly differentiated carcinoma.
* Unidimensionally measurable disease (RECIST criteria).
* ECOG performance status of 0-2
* In the second stage of the study, therapy will be administered with a curative intent and patients should not have recurrent disease or distant metastasis.
* Primary tumor and/or lymphadenopathy should be technically suitable for intratumoral injections. The Otolaryngologist specialist on the head and neck team will determine this feasibility.
* Participating patients should agree to undergo a tumor biopsy at baseline as well as approximately 2 weeks later as specified in study schema.
* Prior treatment
* First stage: any prior treatment, except prior therapy, which specifically and directly targets the EGFR pathway, administered within the last 6 months. No prior radiation therapy to the head and neck.
* Second stage: no prior chemotherapy, biologic/molecular targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer.
* Prior surgical therapy will consist only of incisional or excisional biopsy, including tonsillectomy, and organ sparing procedures, including neck dissection. Any non-biopsy surgical procedure for head and neck cancer must have taken place at least one month before initiating protocol treatment, at the treating physician's discretion.
* Patients must have organ and marrow function as defined below:

Absolute neutrophil count above/equal to 1,000/µL Platelets above/equal to 75,000/µL Hemoglobin above/ equal to 10 g/dL Total bilirubin <2 x upper normal institutional limits Creatinine clearance > 20 mL/min

* Age 18 years or older
* Because radiation therapy is known to be teratogenic and EFGR inhibitors may have teratogenic potential, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation, and for 3 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Severe renal insufficiency (creatinine clearance < 20 mL/min)
* Treatment with anticoagulants, except when used to maintain the patency of a central venous line, or INR >1.5, or PTT ratio >1.5.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements. Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure.
* Patients may not be receiving any other investigational agents.
* No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, DCIS or LCIS of the breast, localized early stage prostate cancer, or malignancy that has been treated with a curative intent with a 3-year disease-free survival.
* Pregnant women are excluded from this study because cetuximab, EGFR AS, and radiation have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cetuximab and EGFR AS, breastfeeding should be discontinued if the mother is treated with cetuximab. The effects of cetuximab and EGFR AS on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with cetuximab. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated. HIV status of the patient will be obtained from the patient's history via discussion with the investigator. HIV testing is not required.
* Prior severe infusion reaction to a monoclonal antibody.
* Patients who are not informed of and are not willing to comply with the investigational nature of the study and have not signed a written informed consent in accordance with institutional and good clinical practice guidelines.
* Phase 2 ONLY (second stage) - Subjects M1 disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Karnad, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at two sites, University of Pittsburgh and University of Texas Health Science Center, San Antonio. Participants were followed to completion of treatment and then long-term follow up.
Pre-assignment Details: Subjects met eligibility for chemotherapy, radiation therapy, and anti-sense DNA injections per protocol
Period: Treatment Period
Arm/Group | EGFR Antisense DNA
Started | 6
Completed | 6
Not Completed | 0
Period: Long-term Follow-up
Arm/Group | EGFR Antisense DNA
Started | 6
Completed | 5
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | EGFR Antisense DNA
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: Years] | 66.5 [50 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 5
  Hispanic or Latino | 4
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Rate
Description: This is a 2-stage clinical trial. In the first stage, toxicity will be the primary endpoint. Toxicity measures will be graded according to NCI CTCAE version 4.0. All AEs reported are grade 1 to grade 3 AEs.
Time Frame: 1 year
Population: Advanced stage squamous cell carcinoma of the head and neck
Measure: Number; unit: Number of adverse events
Arm/Group | EGFR Antisense DNA
Number analyzed (Participants) | 6
Number of adverse events | 20

2. Primary Outcome: Locoregional Progression-free Survival
Description: In the second stage (phase II component), the primary endpoint will be locoregional progression-free survival (PFS) at 1 year measured from patient initial date of treatment to date of documented progression or date of death (in absence of progression).
Time Frame: 1 year
Population: Advanced stage squamous cell carcinoma head and neck.
Measure: Count of Participants; unit: Participants
Arm/Group | EGFR Antisense DNA
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Tumor Response
Description: Clinical secondary endpoints include objective response rates, estimated by the proportion of patients with a best response of complete response (CR), partial response (PR), or stable disease (SD) by RECIST criteria, with corresponding exact 90% confidence limits.
Time Frame: 5 years
Population: No analysis of data was performed since there were not sufficient participants enrolled to provide meaningful results. 11 subjects would have had to complete Phase 1 in order to provide meaningful data for analysis.
Arm/Group | EGFR Antisense DNA
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) will be measured from initial date of treatment to date of documented progression or date of death (in absence of progression) and estimated by the Kaplan-Meier method with 90% confidence limits.
Time Frame: 8 years and 10 months
Population: No data analysis was performed since the study closed early due to low enrollment numbers. There was not sufficient data in order to complete the phase 1 analysis, since 11 subjects would have been required to complete.
Arm/Group | EGFR Antisense DNA
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) will be measured from initial date of treatment to recorded date of death and will be estimated by the Kaplan-Meier method with 90% confidence limits.
Time Frame: 5 years
Population: Advanced stage squamous cell carcinoma head and neck
Measure: Count of Participants; unit: Participants
Arm/Group | EGFR Antisense DNA
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 5 years
Description: Does not differ from clinical trials.gov
Arm/Group | EGFR Antisense DNA
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | EGFR Antisense DNA (N=6)
Hyperglycemia (Endocrine disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Dysguesia (Gastrointestinal disorders) | 3 (3) — Distortion of taste
Odynphagia (Gastrointestinal disorders) | 3/3 (3) — Painful swallowing
Neck burns (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Parotiditis (General disorders) | 1 (1) — Inflammation of parotid gland
Submadibular duct infection (Infections and infestations) | 1 (1) — Infection of a duct situated below the jaw
Hot Flashes/sweats (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bleeding nose
Extremity tremors (Nervous system disorders) | 1 (1)
Skin burns (Skin and subcutaneous tissue disorders) | 1 (1)
Dysnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Difficult or labored breathing
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) — Difficulty swallowing
Peripheral neuropathy (Nervous system disorders) | 1 (1) — Numbness, tingling or muscle weakness in the limb(s)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) — Lower than normal lymphocytes (a type of white blood cells)
Kidney disease (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT01592721/Prot_SAP_000.pdf